CLINICAL TRIAL: NCT04277936
Title: Pharmacologic Modulation of Hippocampal Activity in Psychosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was redesigned and submitted as a new protocol (NCT04559529).
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Stephan Heckers, Department Chair, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VEPP_200218
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Schizophrenia; Psychosis
Keywords: Hippocampus
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Levetiracetam (LEV) 500 mg (Experimental): Participants will take their first dose of 500 mg LEV. After a two hour time window, the participants will complete MRI study. After MRI, patients will begin a 2-week intervention with 250 mg BID oral LEV.
  Interventions: Drug: Levetiracetam 500 mg

INTERVENTIONS:
Drug: Levetiracetam 500 mg — Levetiracetam (LEV) regulates neuronal synaptic exocytosis and calcium-induced neurotransmitter release and has a therapeutic effect on the excitation-inhibition balance of the hippocampus.
  Other Names: Keppra

SUMMARY:
The purpose of this study is to test whether administration of levetiracetam (LEV), a commonly used anti-epileptic that alters neurotransmitter release, can reduce hippocampal hyperactivity. Specifically, we will utilize two functional magnetic resonance imaging (MRI) techniques: 1) blood oxygen level dependence (BOLD) contrast will assess activity with a visual scene processing task that engages the anterior hippocampus and 2) arterial spin labeling (ASL) will assess baseline activity. This study will also assess whether patients have improvement in their symptoms after receiving LEV. Previous studies in people with psychotic disorders have shown that the hippocampus is hyperactive and more activity correlates with worsening of clinical symptoms. Therefore, the aim of this study is to use an intervention to further understand the underlying mechanisms of the hippocampus in psychosis.

ELIGIBILITY:
Inclusion criteria for psychosis subjects:

1. Men and women age 18 - 65.
2. Communicative in English.
3. Provide voluntary, written informed consent.
4. Physically healthy by medical history.
5. BMI > 17.5 and < 45.
6. Diagnosis of a psychotic disorder confirmed by Structured Clinical Interview for DSM-V (SCID) or diagnostic interview with a trained clinician.
7. Stable medication regimen over at least the past two weeks, including the use of either an oral or intramuscular administration of an antipsychotic medication.
8. For females, no longer of child-bearing potential, or agreeing to practice effective contraception during the study; and,
9. For females of child-bearing potential, must have negative urine pregnancy test at time of screening visit and before each testing day.
10. Not breastfeeding/nursing at time of screening or at any time during the study.

Inclusion criteria for healthy controls All of the above except for subjects will be psychiatrically healthy and not taking psychotropic or potentially psychoactive prescription medication.

Exclusion criteria for psychosis subjects

1. Age less than 18 or greater than 65.
2. Not communicative in English.
3. Unable to provide written informed consent.
4. Current medical or neurological illness.
5. History of severe head trauma.
6. BMI < 17.5 or > 45.
7. Meets criteria for diagnosis of substance or alcohol use disorder within the past month.
8. Positive urine pregnancy test at time of screening, before each testing day, or any potential concern for pregnancy at any time during the study.
9. Breastfeeding/nursing at time of screening or at any time during the study.
10. Conditions that preclude MR scanning
11. Conditions that preclude study drug administration

Exclusion criteria for healthy controls

All of the above and in addition:

1. Current use of psychotropic or potentially psychoactive prescription medication.
2. Major psychiatric disorder as determined by DSM-V (major depression, bipolar disorder, obsessive compulsive disorder, post-traumatic stress disorder, etc)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levetiracetam (LEV) 500 mg
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Data were collected for a single subject, but study design was changed and study was discontinued. No data were analyzed.
Arm/Group | Levetiracetam (LEV) 500 mg
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Hippocampal Activity (Arterial Spin Labeling [ASL] Study)
Description: Change in ASL signal after drug administration
Time Frame: 2 hours and 2 weeks after administration
Population: Data were collected for a single subject, but study design was changed and study was discontinued.
Arm/Group | Levetiracetam (LEV) 500 mg
Number analyzed (Participants) | 0

2. Primary Outcome: Hippocampal Recruitment (BOLD Study)
Description: Change in BOLD signal after drug administration
Time Frame: 2 hours and 2 weeks after administration
Population: Data were collected for a single subject, but study design was changed and study was discontinued.
Arm/Group | Levetiracetam (LEV) 500 mg
Number analyzed (Participants) | 0

3. Secondary Outcome: Cognitive Symptoms
Description: Change in eye-tracking relational memory task
Time Frame: 2 weeks after administration
Population: No data were collected.
Arm/Group | Levetiracetam (LEV) 500 mg
Number analyzed (Participants) | 0

4. Secondary Outcome: Positive and Negative Symptoms
Description: Change PANSS score
Time Frame: 2 weeks after administration
Population: Healthy participant; outcome measure does not apply
Arm/Group | Levetiracetam (LEV) 500 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 weeks The protocol is: a) single dose of 500mg LEV, b) neuroimaging session #1, c) 500mg LEV for 2-weeks and d) imaging session #2. This participant only took a single 500mg dose and never advanced to the protocol components c) and d), i.e. did not complete the study protocol. 93% of LEV is cleared in 48 hours, so monitoring is not necessary beyond 1 week.
Description: no adverse events
Arm/Group | Levetiracetam (LEV) 500 mg
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT04277936/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT04277936/ICF_001.pdf